CLINICAL TRIAL: NCT01783119
Title: Effect of Aloe Vera in the Inflammation of Patients With Mild Ulcerative Colitis
Acronym: AVIUC
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Medical Sciences and Nutrition, Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Jesús Kazuo Yamamoto Furusho, MD PhD, National Institute of Medical Sciences and Nutrition, Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REF.589
Record Dates: First submitted 2013-01-31; First posted 2013-02-04 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-01

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; Aloe Vera
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aloe Vera (Experimental): Consume 200 ml of aloe vera gel per day over a period of three months
  Interventions: Dietary Supplement: Aloe Barbadensis Miller
- water (Placebo Comparator): Consume 200 ml of placebo per day over a period of three months
  Interventions: Dietary Supplement: placebo water

INTERVENTIONS:
Dietary Supplement: Aloe Barbadensis Miller
  Arms: Aloe Vera
Dietary Supplement: placebo water
  Arms: water

SUMMARY:
The Ulcerative Colitis (UC) belongs to the group of diseases called Inflammatory Bowel Disease (IBD) which is characterized by a chronic ulceration of the colon. The conventional treatment can have adverse effects and does not guarantee effectiveness in some patients requiring aggressive therapy using adjuvant therapy Aloe vera has been shown to have a beneficial effect in different disease, and have an anti-inflammatory effect in UC patients. Objective: Measuring the effect of the consumption of 200 ml of aloe vera gel daily for a period of three months, in the degree of inflammation in patients with mild UC based on Mayo scale and quantification of IL-6 in the colonic mucosa.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis by histopathology of Ulcerative Colitis with mild activity level clinical, Endoscopic and histological.
* Extent of disease: pancolitis, ulcerative proctitis and left.
* Being treated with 5 - aminosalicylates (5-ASA).
* Belonging to the National Institute of Medical Sciences and Nutrition "Salvador Zubirán".
* Signed informed consent.

Exclusion Criteria:

* Autoimmune diseases (lupus, HIV, cancer and any hepatitis).
* Another type of colitis (indeterminate, infectious drug and Crohn's Disease.
* Previous total colectomy.
* Body mass index less than 19.9 kg/m2 or greater than 40 kg/m2.
* Patients in remission histology, clinical and endoscopic.
* Under treatment with steroids, azathioprine, diuretics and anticoagulants.
* Use Aloe Vera or some natural therapy.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Full Mayo Score | 3 months
Interleukine - 6 | 3 months
  Quantification in mucosal Biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Jesús K Yamamoto-Furusho, MD, PhD, Study Chair — INCMNSZ; Lizzette C Alfaro, Principal Investigator — INCMNSZ
Locations (1):
- National Institute of Medical Science and Nutrition, Salvador Zubirán, D.f., Tlalpan, Mexico

REFERENCES:
- [Background] Molodecky NA, Soon IS, Rabi DM, Ghali WA, Ferris M, Chernoff G, Benchimol EI, Panaccione R, Ghosh S, Barkema HW, Kaplan GG. Increasing incidence and prevalence of the inflammatory bowel diseases with time, based on systematic review. Gastroenterology. 2012 Jan;142(1):46-54.e42; quiz e30. doi: 10.1053/j.gastro.2011.10.001. Epub 2011 Oct 14. PMID 22001864
- [Background] Bosques-Padilla FJ, Sandoval-Garcia ER, Martinez-Vazquez MA, Garza-Gonzalez E, Maldonado-Garza HJ. [Epidemiology and clinical characteristics of ulcerative colitis in north-eastern Mexico]. Rev Gastroenterol Mex. 2011 Jan-Mar;76(1):34-8. Spanish. PMID 21592901
- [Background] Sanjurjo-García, J. L., Aranda-Jiménez, G., Garuño-Delgado, R., y García-Manzo, N. T. Guías clínicas de diagnóstico y tratamiento de la colitis ulcerativa crónica idiopática (CUCI). Diagnóstico. Utilidad de los datos clínicos y análisis de laboratorio.Rev. Gastroenterol Mex. 2007; 72(2):136-138.
- [Background] López-Rosés L, Olivencia-Palomar P. Colonoscopia. Rev. esp. enferm. dig. 100(6): 372-372; 2008.
- [Background] Martinez-Benitez, B. Características morfológicas de la enfermedad intestinal inflamatoria idiopática. En: Yamamoto-Furusho, JK. Enfermedad Inflamatoria Intestinal: Aspectos básicos y clínicos.2010; México, D.F: Alfil
- [Background] Villeda-Ramirez M.A. Etiopatogenia de la enfermedad inflamatoria intestinal. En: Yamamoto-Furusho, JK.. Enfermedad Inflamatoria Intestinal: Aspectos básicos y clínicos. 2010; México, D.F: Alfil
- [Background] World Healh Organization. National policy on traditional medicine and regulation of herbal medicines .Report of a WHO global survey. Geneve 2005
- [Background] Wild GE, Drozdowski L, Tartaglia C, Clandinin MT, Thomson AB. Nutritional modulation of the inflammatory response in inflammatory bowel disease--from the molecular to the integrative to the clinical. World J Gastroenterol. 2007 Jan 7;13(1):1-7. doi: 10.3748/wjg.v13.i1.1. PMID 17206749
- [Background] Atherton P. Aloe vera revisited. British Journal of Phytotherapy 1998; 4(4): 176-183.
- [Background] Holdsworth DK. Chromones in aloe species. I. Aloesin--a C-glucosyl-7-hydroxychromone. Planta Med. 1971 Apr;19(4):322-5. doi: 10.1055/s-0028-1099649. No abstract available. PMID 5573544
- [Background] Siddharthan K. Health insurance coverage of the immigrant elderly. Inquiry. 1991 Winter;28(4):403-12. PMID 1761313
- [Background] Avila H, Rivero J, Herrera F, Fraile G. Cytotoxicity of a low molecular weight fraction from Aloe vera (Aloe barbadensis Miller) gel. Toxicon. 1997 Sep;35(9):1423-30. doi: 10.1016/s0041-0101(97)00020-2. PMID 9403965
- [Background] Curciarello J, De Ortuzar S, Borzi S, Bosia D. [Severe acute hepatitis associated with intake of Aloe vera tea]. Gastroenterol Hepatol. 2008 Aug-Sep;31(7):436-8. doi: 10.1157/13125590. Spanish. PMID 18783689
- [Background] Bottenberg MM, Wall GC, Harvey RL, Habib S. Oral aloe vera-induced hepatitis. Ann Pharmacother. 2007 Oct;41(10):1740-3. doi: 10.1345/aph.1K132. Epub 2007 Aug 28. PMID 17726067
- [Background] Rabe C, Musch A, Schirmacher P, Kruis W, Hoffmann R. Acute hepatitis induced by an Aloe vera preparation: a case report. World J Gastroenterol. 2005 Jan 14;11(2):303-4. doi: 10.3748/wjg.v11.i2.303. PMID 15633238
- [Background] El-Shemy HA, Aboul-Soud MA, Nassr-Allah AA, Aboul-Enein KM, Kabash A, Yagi A. Antitumor properties and modulation of antioxidant enzymes' activity by Aloe vera leaf active principles isolated via supercritical carbon dioxide extraction. Curr Med Chem. 2010;17(2):129-38. doi: 10.2174/092986710790112620. PMID 19941474
- [Background] Kim K, Kim H, Kwon J, Lee S, Kong H, Im SA, Lee YH, Lee YR, Oh ST, Jo TH, Park YI, Lee CK, Kim K. Hypoglycemic and hypolipidemic effects of processed Aloe vera gel in a mouse model of non-insulin-dependent diabetes mellitus. Phytomedicine. 2009 Sep;16(9):856-63. doi: 10.1016/j.phymed.2009.02.014. Epub 2009 Mar 19. PMID 19303272
- [Background] Davis RH, Donato JJ, Hartman GM, Haas RC. Anti-inflammatory and wound healing activity of a growth substance in Aloe vera. J Am Podiatr Med Assoc. 1994 Feb;84(2):77-81. doi: 10.7547/87507315-84-2-77. PMID 8169808
- [Background] Davis RH, Leitner MG, Russo JM, et al. Biological activity of Aloe vera. Med Sci Res ; 15: 235, 1987b.
- [Background] Guo J, Xiao B, Zhang S, Liu D, Liao Y, Sun Q. Growth inhibitory effects of gastric cancer cells with an increase in S phase and alkaline phosphatase activity repression by aloe-emodin. Cancer Biol Ther. 2007 Jan;6(1):85-8. doi: 10.4161/cbt.6.1.3553. PMID 17172820
- [Background] Stochastic ESR analysis of rat liver and hepatoma mitochondrial lipids. Biophys Struct Mech. 1978 Apr 13;4(2):111-4. doi: 10.1007/BF00539225. PMID 206295
- [Background] Hatano T, Kusuda M, Inada K, Ogawa TO, Shiota S, Tsuchiya T, Yoshida T. Effects of tannins and related polyphenols on methicillin-resistant Staphylococcus aureus. Phytochemistry. 2005 Sep;66(17):2047-55. doi: 10.1016/j.phytochem.2005.01.013. PMID 16153408
- [Background] Saccu D, Bogoni P, Procida G. Aloe exudate: characterization by reversed phase HPLC and headspace GC-MS. J Agric Food Chem. 2001 Oct;49(10):4526-30. doi: 10.1021/jf010179c. PMID 11599983
- [Background] Speranza G, Morelli CF, Tubaro A, Altinier G, Duri L, Manitto P. Aloeresin I, an anti-inflammatory 5-methylchromone from cape aloe. Planta Med. 2005 Jan;71(1):79-81. doi: 10.1055/s-2005-837756. PMID 15678379
- [Background] León Sarabia JE, Rosales Clares V, Rosales Clares RA. Alternativas terapéuticas para pacientes portadores de colitis idiopática utilizando aloe vera l. (sábila). Una experiencia. REV CUBANA PLANT MED.3(3):102-5,1999.
- [Background] Langmead L, Makins RJ, Rampton DS. Anti-inflammatory effects of aloe vera gel in human colorectal mucosa in vitro. Aliment Pharmacol Ther. 2004 Mar 1;19(5):521-7. doi: 10.1111/j.1365-2036.2004.01874.x. PMID 14987320
- [Result] Gower-Rousseau C, Salomez JL, Dupas JL, Marti R, Nuttens MC, Votte A, Lemahieu M, Lemaire B, Colombel JF, Cortot A. Incidence of inflammatory bowel disease in northern France (1988-1990). Gut. 1994 Oct;35(10):1433-8. doi: 10.1136/gut.35.10.1433. PMID 7959201
- [Result] Yamamoto-Furusho JK. Clinical epidemiology of ulcerative colitis in Mexico: a single hospital-based study in a 20-year period (1987-2006). J Clin Gastroenterol. 2009 Mar;43(3):221-4. doi: 10.1097/MCG.0b013e31817a76b4. PMID 19057395
- [Result] Knigge KL. Inflammatory bowel disease. Clin Cornerstone. 2002;4(4):49-60. doi: 10.1016/s1098-3597(02)90005-0. PMID 12739326
- [Result] Yamamoto-Furusho ,JK, Villalobos, JJ, Olvera, MA, Valdovinos, MA. Colitis ulcerosa crónica inespecífica (CUCI). Gastroenterología. 59. México, Ed. Méndez. 2006; 401-4.
- [Result] Bousoño C, Ramos E. Enfermedad Inflamatoria Intestinal. Bol Pediatr 46 (1): 91-99, 2006.
- [Result] Baumgart DC, Sandborn WJ. Inflammatory bowel disease: clinical aspects and established and evolving therapies. Lancet. 2007 May 12;369(9573):1641-57. doi: 10.1016/S0140-6736(07)60751-X. PMID 17499606
- [Result] Feagan BG, Greenberg GR, Wild G, Fedorak RN, Pare P, McDonald JW, Dube R, Cohen A, Steinhart AH, Landau S, Aguzzi RA, Fox IH, Vandervoort MK. Treatment of ulcerative colitis with a humanized antibody to the alpha4beta7 integrin. N Engl J Med. 2005 Jun 16;352(24):2499-507. doi: 10.1056/NEJMoa042982. PMID 15958805
- [Result] Podolsky DK. Inflammatory bowel disease. N Engl J Med. 2002 Aug 8;347(6):417-29. doi: 10.1056/NEJMra020831. No abstract available. PMID 12167685
- [Result] Fonseca-Camarillo GC, Villeda-Ramirez MA, Sanchez-Munoz F, Barreto-Zuniga R, Dominguez-Lopez A, Uribe-Esquivel M, Yamamoto-Furusho JK. [IL-6 and TNF-alpha gene expression in the rectal mucosal of patients with chronic idiopathic ulcerative colitis and controls]. Rev Gastroenterol Mex. 2009 Oct-Dec;74(4):334-40. Spanish. PMID 20423763
- [Result] Mane Almero J. [In vivo experimental models of inflammatory bowel disease and colorectal cancer]. Nutr Hosp. 2007 Mar-Apr;22(2):178-89. Spanish. PMID 17416034
- [Result] Blonski W, Buchner AM, Lichtenstein GR. Inflammatory bowel disease therapy: current state-of-the-art. Curr Opin Gastroenterol. 2011 Jul;27(4):346-57. doi: 10.1097/MOG.0b013e328347aef3. PMID 21654383
- [Result] Park MY, Kwon HJ, Sung MK. Intestinal absorption of aloin, aloe-emodin, and aloesin; A comparative study using two in vitro absorption models. Nutr Res Pract. 2009 Spring;3(1):9-14. doi: 10.4162/nrp.2009.3.1.9. Epub 2009 Mar 31. PMID 20016696